CLINICAL TRIAL: NCT01521182
Title: Effect of the Consumption of a Fermented Dairy Drink on the Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: NU356
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Free-living Elderly
Keywords: Probiotic - dairy product - influenza vaccination - healthy elderly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 = Tested product (Active Comparator)
  Interventions: Other: 1-Fermented Dairy Product (test)
- 2 = Control product (Placebo Comparator)
  Interventions: Other: 2-Milk-based non-fermented dairy product (control)

INTERVENTIONS:
Other: 1-Fermented Dairy Product (test) — 1 = Intervention 1 (test product)
  Arms: 1 = Tested product
Other: 2-Milk-based non-fermented dairy product (control) — 2 = Intervention 2 (control product)
  Arms: 2 = Control product

SUMMARY:
The purpose of this study is to determine whether the regular consumption of the active product enhances the immune function, in comparison to the control product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy free-living both gender elderly aged from 65 to 80 years old on the day of inclusion
* Able to comply with all the trial procedures
* Having given written consent to take part in the study prior to participation.
* Body mass index (BMI): 18,5 < BMI < 30 kg/m².

Exclusion Criteria:

* Contra-indication to any of the products and procedures used for the study purpose
* Participation in another clinical trial
* People currently institutionalised
* Immunocompromised conditions or other conditions that may impact the immune response or the product effect
* Subjects suffering from a not stabilized chronic disease
* Subjects suffering from a sever acute or chronic disease
* Subjects suffering from a condition which is at a stage where it might prevent him/her from being able or willing to comply with the study procedures or completion
* Subject known to be deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Subject identified as employees of the Investigator or study centre, with direct involvement in the proposed study or other studies under the direction of that Investigator or study centre, as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the centre's employees or the Investigator.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 550 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Centre for the Evaluation of Vaccination, Vaccine & Infectious Disease Institute - University of Antwerp, Wilrijk - Antwerp, Belgium